CLINICAL TRIAL: NCT02296736
Title: The Pre-operative Pathway in Pancreatic Head Malignancy-assessment of the Diagnostic Accuracy of Staging CT Scan
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/P/090; 14/SC/1391 PR (Other: National Research Ethics Service (NRES))
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Cancer of Pancreas
Keywords: computerised tomography (CT) scan; diagnostic accuracy; Pancreatic head malignancy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic malignancy: All patients who have undergone surgery for presumed pancreatic malignancy in Derriford Hospital between Jan 2006 and Jan 14 and had a Computerised tomography (CT) scan.
  Interventions: Radiation: Computerised tomography (CT) scan

INTERVENTIONS:
Radiation: Computerised tomography (CT) scan — Retrospective review of CT scans

SUMMARY:
Our aim is to assess the ability of scans to distinguish the organ of origin of pancreatic head malignant tumours and to predict the resectability based on the preoperative imaging. To achieve this, a retrospective review of the preoperative CT scans will be conducted for all patients with pancreatic head malignancy treated at the Peninsula Hepato-Pancreatico-Biliary (HPB) cancer unit between January 2006 till January 2014.

DETAILED DESCRIPTION:
Pancreatic cancer arises from the glandular part of the pancreas and is the fifth most common cause for cancer related death in the UK. It. Ampullary carcinoma arises from the epithelium of the ampulla of Vater into which the common bile duct and pancreatic duct drain. Cholangiocarcinoma arises from the bile duct epithelium, and may occur within the intra-pancreatic portion of the distal common bile duct mimicking a pancreatic malignancy. Cancers arising from these origins often cause obstructive jaundice and are hard to distinguish. Surgery is indicated for the treatment of these types of malignant tumours, and the definitive final diagnosis is usually not known until the specimen is examined. This situation does not allow specific treatment to be given pre-operatively, so-called 'neo-adjuvant therapy'. The rationale for this approach is that in a proportion of patients the tumour will be made smaller by this treatment, which may facilitate surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone surgery for presumed pancreatic malignancy in Derriford Hospital between Jan 2006 and Jan 14 will be included.

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective review of imaging of all patients who have undergone surgery for presumed pancreatic malignancy in Derriford Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Review pre-operative imaging to distinguish the organ of origin of pancreatic head tumours | 8 years
  Retrospective review of imaging of patients who have undergone surgery for presumed pancreatic malignancy

SECONDARY OUTCOMES:
Resectabilty of the pancreatic tumour | 8 years
  Retrospective review of imaging of patients who have undergone surgery for presumed pancreatic malignancy

CONTACTS AND LOCATIONS:
Overall Officials: David Stell, MBBS, PhD, Study Director — University Hospital Plymouth NHS Trust; Bassem Amr, MBBS, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom

REFERENCES:
- [Derived] Amr B, Shahtahmassebi G, Aroori S, Bowles MJ, Briggs CD, Stell DA. Variation in survival after surgery for peri-ampullary cancer in a regional cancer network. BMC Surg. 2017 Mar 7;17(1):23. doi: 10.1186/s12893-017-0220-3. PMID 28270136